CLINICAL TRIAL: NCT01226862
Title: Advancing Telestroke Care: A Prospective Observational Study
Acronym: ATC
Status: Completed | Type: Observational
Sponsor: National Stroke Association, United States (Other)
Collaborators: University of Southern California (Other); Mayo Clinic (Other); Swedish Medical Center (Other); University of Utah (Other); California Pacific Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NSA Telestroke
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Stroke
Keywords: Stroke; Telemedicine; Telestroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hub Hospital: Hub Hospital Cohort: Joint Commission-certified Primary Stroke Centers where patients are treated using hospital-based stroke teams and pathways; these hospital personnel also provide telemedicine consultation to satellite hospitals.
- Spoke Hospital: Spoke Hospital Cohort: non-stroke center certified sites, where patients are treated at an in-network telestroke community hospital using telemedicine technology with consultation provided by physicians from a hub hospital.
- Control Hospital: Control Hospital Cohort: non-stroke center certified sites with no telemedicine services.

SUMMARY:
This study will promote the development and economic sustainability of telemedicine for acute stroke treatment.

DETAILED DESCRIPTION:
The goal of this study is to promote the development and economic sustainability of telemedicine for acute stroke treatment. The study's objectives are 1) to determine if the use of telemedicine consultations for stroke patients will improve their care per guidelines compared to stroke patients treated by control hospitals; and 2) to determine if the care per guidelines provided via telemedicine consultations for stroke patients will be similar or equivalent to care per guidelines provided to stroke patients treated at hub hospitals.

The Advancing Telestroke Care study will establish treatment and outcomes in three distinct study cohorts: hub telemedicine hospital, spoke telemedicine hospital and non-telemedicine control hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Acute ischemic stroke within 12 hours of stroke onset

Exclusion Criteria:

* Life expectancy less than 90 days
* Patient unwilling to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 subjects meeting inclusion and exclusion criteria will be enrolled consecutively over approximately 12 months and followed for 90 days post-stroke.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
IV tPA administration | Day 7/Discharge
  Correctness of decisions regarding IV tPA administration in acute stroke

SECONDARY OUTCOMES:
Multiple Study Assessments | Day 7 and/or Day 30 and/or Day 90 and/or at discharge
  There are 23 assessments, after stroke, for outcome measures. They include: hospital transfers, treatment with reperfusions therapies, treatment with antiplatelets, hypertension treatment, hyperglycemia treatment, hyperlipidemia treatment, symptomatic ICH, mortality, imaging/diagnostic data, stroke and rehab scale scores, number of hospitalizations since last assessment, hospital LOS, discharge location, number of physician visits, and work status.

CONTACTS AND LOCATIONS:
Overall Officials: Gene Sung, MD, MPH, Principal Investigator — University of Southern California, Los Angeles
Locations (1):
- University of Southern California, Los Angeles, California, United States